CLINICAL TRIAL: NCT03756623
Title: Effect of Metformin and Probiotics on Gut Microbiome in Healthy Subjects: a Randomized, Double-blind Study.
Brief Title: Effect of Metformin and Probiotics on Gut Microbiome in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Mingming Zhang, Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: microbiome2018
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drug: Metformin powder (Experimental): 0.5g of Metformin powder administered three times a day orally before meal
  Interventions: Drug: Metformin powder
- Drug: Probiotics powder (Experimental): 0.5g of Probiotics powder administered three times a day orally before meal
  Interventions: Drug: Probiotics powder
- Drug: Placebo powder (Placebo Comparator): 0.5g of Placebo powder administered three times a day orally before meal
  Interventions: Other: Placebo powder

INTERVENTIONS:
Drug: Metformin powder — 0.5g of Metformin powder administered three times a day orally before meal
  Arms: Drug: Metformin powder
Drug: Probiotics powder — 0.5g of Probiotics powder administered three times a day orally before meal
  Arms: Drug: Probiotics powder
Other: Placebo powder — 0.5g of Placebo powder administered three times a day orally before meal
  Arms: Drug: Placebo powder

SUMMARY:
This clinical trial is designed to evaluate the alteration of gut microbiome in healthy subjects after a 12-week metformin and/or probiotics administration.

DETAILED DESCRIPTION:
Gut microbiome dysbiosis have been linked with the onset and progression of several diseases. Metformin and probiotics have been confirmed to function partly by regulating the gut microbiome. The investigators are now wondering if metformin/probiotics treatment will change the gut microbiota in healthy subjects and show some benefits.

In this study, about 60 healthy subjects will be enrolled. Participants will be randomly assigned into one of the following three groups: Metformin powder (0.5g tid po), Probiotics powder (0.5g tid po), Placebo powder (0.5g tid po), for 12 weeks.

Blood and stool samples will be collected before and after treatment. Fasting glucose levels, fasting insulin levels, serum lipid profiles, inflammation markers and alteration of gut microbiota will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Between 20-60 years of age.
2. Healthy subjects without known diseases.

Exclusion Criteria:

1. During pregnancy and lactation period.
2. Impaired liver function, impaired renal function, mental disease, severe infection, severe anemia, severe heart disease and neutropenia disease.
3. Use of metformin/antibiotics within 3 months.
4. Immunodeficient or use of immunosuppressive drugs.
5. Previous history of gastrointestinal surgery or diseases (such as peptic ulcer, irritable bowel syndrome, inflammatory bowel disease or other gastrointestinal disorder).
6. Medical conditions or diseases that may affect subject safety or confound study results in the opinion of the investigator.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Gut microbiota alterations | 12 weeks
  Gut microbiota composition and function will be assessed before and after study.

CONTACTS AND LOCATIONS:
Overall Officials: Mingming Zhang, MD,PhD, Principal Investigator — Drum Tower hospital affiliated to Nanjing University Medical School
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided